CLINICAL TRIAL: NCT03568916
Title: Safety and Effectiveness of Direct Oral Anticoagulants for Stroke Prevention in Non-valvular Atrial Fibrillation: a Multi-database Cohort Study With Meta-analysis (DOACs vs DOACs)
Brief Title: Direct Oral Anticoagulants in Patients With Atrial Fibrillation (DOACs vs DOACs)
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q16-13A
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; Systemic Embolization; Major Bleed; Myocardial Infarction; All-cause Mortality
Keywords: Direct oral anticoagulants; Safety; Atrial fibrillation; Ischemic stroke; Systemic embolization
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Myocardial Infarction | interventions — apixaban; Dabigatran; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rivaroxaban vs dabigatran: Patients diagnosed with non-valvular atrial fibrillation who initiated their oral anticoagulation with rivaroxaban or dabigatran at cohort entry date, and did not have a previous prescription for any oral anticoagulant in the prior year.
  Interventions: Drug: Dabigatran (ATC B01AE07); Drug: Rivaroxaban (ATC B01AF01)
- Apixaban vs dabigatran: Patients diagnosed with non-valvular atrial fibrillation who initiated their oral anticoagulation with apixaban or dabigatran at cohort entry date, and did not have a previous prescription for any oral anticoagulant in the prior year.
  Interventions: Drug: Apixaban (ATC B01AF02); Drug: Dabigatran (ATC B01AE07)
- Apixaban vs rivaroxaban: Patients diagnosed with non-valvular atrial fibrillation who initiated their oral anticoagulation with apixaban or rivaroxaban at cohort entry date, and did not have a previous prescription for any oral anticoagulant in the prior year.
  Interventions: Drug: Apixaban (ATC B01AF02); Drug: Rivaroxaban (ATC B01AF01)

INTERVENTIONS:
Drug: Apixaban (ATC B01AF02) — Exposure to apixaban (ATC B01AF02) will be defined as a new prescription for apixaban at cohort entry date in patients diagnosed with non-valvular atrial fibrillation. Patients are considered exposed until end of follow-up regardless of switch or interruption.
  Other Names: Eliquis
  Groups: Apixaban vs dabigatran; Apixaban vs rivaroxaban
Drug: Dabigatran (ATC B01AE07) — Exposure to dabigatran (ATC B01AE07) will be defined as a new prescription for dabigatran at cohort entry date in patients diagnosed with non-valvular atrial fibrillation. Patients are considered exposed until end of follow-up regardless of switch or interruption.
  Other Names: Pradaxa
  Groups: Apixaban vs dabigatran; Rivaroxaban vs dabigatran
Drug: Rivaroxaban (ATC B01AF01) — Exposure to rivaroxaban (ATC B01AF01) will be defined as a new prescription for rivaroxaban at cohort entry date in patients diagnosed with non-valvular atrial fibrillation. Patients are considered exposed until end of follow-up regardless of switch or interruption.
  Other Names: Xarelto
  Groups: Apixaban vs rivaroxaban; Rivaroxaban vs dabigatran

SUMMARY:
The purpose of this study is to assess safety and effectiveness of direct oral anticoagulants (DOACs) for stroke prevention in patients with non-valvular atrial fibrillation (AF). The comparison of DOACs between themselves is of interest.

The investigators will carry out separate population-based, matched cohort studies, using health administrative databases in nine jurisdictions in Canada, the UK and the US. New users of DOACs for stroke prevention in non-valvular AF will be eligible to enter the cohorts. Follow-up will continue until a hospitalization or emergency department visit for a stroke. The results from the separate sites will be combined by meta-analysis to provide an overall assessment of the safety and effectiveness of the different anticoagulation regimens in stroke prevention in AF.

The investigators hypothesize that different DOACs will have similar safety and effectiveness profiles.

DETAILED DESCRIPTION:
The objective of this study is to assess safety and effectiveness of direct oral anticoagulants (DOACs) for stroke prevention in patients with non-valvular atrial fibrillation (AF).

A common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from nine jurisdictions (the Canadian provinces of Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, Saskatchewan, as well as the United Kingdom (UK) Clinical Practice Research Datalink (CPRD) and the United States (US) Marketscan). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. The data in Alberta, Nova Scotia, and Ontario will be restricted to patients aged 65 years and older, as prescription data are not available for younger patients. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data. US MarketScan includes individuals and their dependents covered by large US employer health insurance plans, and government and public organizations.

In each jurisdiction, the investigators will assemble a base cohort that includes all patients newly prescribed a DOAC for stroke prevention in AF. Study period will be from the date of the first DOAC approval for stroke prevention in AF at each site to the date of latest data availability at each site. All patients newly dispensed a DOAC (i.e. with no prescription for any oral anticoagulant in the prior year) with a diagnosis of AF within the 3 years prior to the date of the prescription will be eligible to be included into the study cohorts, given they present no exclusion criteria. The date of study cohort entry will be defined by the prescription (for CPRD) or dispensation (for all other sites) date of the newly prescribed DOAC. Patients will be censored at the earliest of death, end of healthcare coverage, or the end of the study period, whichever occurs first.

Exposure to a DOAC will be defined as a new prescription for a DOAC (apixaban, dabigatran, rivaroxaban) on the date of cohort entry. The investigators will use an analysis analogous to an intention-to-treat approach. The primary outcome will be defined as a hospitalization or emergency department visit for ischemic stroke or systemic embolization. The secondary outcomes will be: 1) major bleeding; 2) a composite of stroke (ischemic or hemorrhagic), systemic embolization, major bleeding or all-cause mortality; 3) myocardial infarction; 4) gastrointestinal bleeding; 5) intracranial bleeding; and 6) all-cause mortality.

The study cohort will be analyzed using a matched cohort design. In each participating site, three distinct study cohorts will be assembled, one for each of the following comparisons, nested in the same base cohort: 1) dabigatran vs. rivaroxaban, 2) dabigatran vs. apixaban, and 3) rivaroxaban vs. apixaban. DOAC users will be matched 1:1 to DOAC users on sex, age, cohort entry date, and propensity score (which will be constructed using a multivariable logistic regression model estimating the odds of being treated with DOACs, while adjusting for a number of pre-identified covariates to account for baseline differences at the time of cohort entry). Cox-proportional hazards regression models will be used to estimate adjusted hazards ratios (HRs) and corresponding 95% confidence intervals (CIs) for ischemic stroke or systemic embolization in the three cohorts. Meta-analyses of the site-specific results will be performed using random effects models. As secondary analyses, the composite outcome will be stratified by age (<85 and ≥85) and sex. In addition, an as treated analysis using inverse probability of censoring weights (IPCW) will be performed to account for non-random censoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new prescription for an oral anticoagulant that had a diagnosis of atrial fibrillation or atrial flutter within the 3 years prior to the date of the prescription
* Patients aged 18 years or older (except Alberta, Nova Scotia, and Ontario, where patients will be aged at least 66 years or older)

Exclusion Criteria:

* Patients with less than one year of data availability prior to cohort entry
* Patients with a diagnosis of valvular disease (including rheumatic heart disease) or prior cardiac valve surgery
* Patients with a diagnosis of venous thromboembolic disease in the year prior to cohort entry
* Patients who underwent hemodialysis in the 90 days prior to cohort entry
* Patients with a hip, femur, or knee surgery in the 30 days prior to cohort entry
* Patients with a diagnosis of antiphospholipid syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients newly anticoagulated from the date of the first DOAC approval for stroke prevention in AF (in each site) to the date of the latest data availability at each site, that had a diagnosis of AF within the 3 years prior to the date of the prescription.
Sampling Method: Probability Sample
Enrollment: 227579 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Ischemic stroke (IS) or systemic embolization (SE) | Patients will be followed from date of first DOAC prescription (cohort entry date) until a hospitalization or emergency department visit for IS or SE, censoring due to death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
  Patients hospitalized or visiting the emergency department for a stroke or a systemic embolization recorded as the most responsible diagnosis in either the discharge abstract or hospitalization record with the following ICD codes:
  Ischemic stroke:
  ICD-9 codes: 434.x ICD-10 codes: I63.x, I64.x
  Systemic embolization:
  ICD-9 codes: 444.x ICD-10 codes: I74.x

SECONDARY OUTCOMES:
Major bleeding | Patients will be followed from date of first DOAC prescription (cohort entry date) until a hospitalization or emergency department visit for major bleed, censoring due to death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
  Patients hospitalized or visiting the ER for a major bleed composite recorded as the most responsible diagnosis in either the discharge abstract or hospitalization record with the following ICD codes:
  Intracranial bleeding (including hemorrhagic stroke):
  ICD-9 codes: 430.x, 431.x, 432.x ICD-10 codes: I60.x, I61.x, I62.x
  Gastrointestinal bleeding:
  ICD-9 codes: 456.0, 531.0, 531.2, 531.4, 531.6, 532.0, 532.2, 532.4, 532.6, 533.0, 533.2, 533.4, 533.6, 534.0, 534.2, 534.4, 534.6, 569.3, 578.x ICD-10 codes: I85.0, I98.3, K25.0, K25.2, K25.4, K25.6, K26.0, K26.2, K26.4, K26.6, K27.0, K27.2, K27.4, K27.6, K28.0, K28.2, K28.4, K28.6, K29.0, K55.21, K62.5, K63.81, K92.0, K92.1, K92.2
  Ocular bleeding:
  ICD-9 codes: 362.81, 363.6x, 376.32, 379.23, 377.42 ICD-10 codes: H31.3, H35.6, H43.1, H45.0
  Other bleeding causing ER visit or hospitalization:
  ICD-9 codes: 459.0, 596.7, 599.7, 627.1, 719.1, 729.92, 784.7, 784.8, 786.3 ICD-10 codes: D68.3, K66.1, M25.0x, N02.x
All-cause mortality | Patients will be followed from date of first DOAC prescription (cohort entry date) until death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
Myocardial infarction | Patients will be followed from date of first DOAC prescription (cohort entry date) until a hospitalization for a myocardial infarction, censoring due to death, end of healthcare coverage, or for up to 65 months, whichever occurs first.
  Patients hospitalized for a myocardial infarction recorded as the most responsible diagnosis in hospitalization record with the following ICD codes:
  ICD-9 code: 410.x ICD-10 code: I21.x

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Durand, MD, MSc, FRCPC, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Durand M, Schnitzer ME, Pang M, Carney G, Eltonsy S, Filion KB, Fisher A, Jun M, Kuo IF, Matteau A, Paterson JM, Quail J, Renoux C; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Effectiveness and safety among direct oral anticoagulants in nonvalvular atrial fibrillation: A multi-database cohort study with meta-analysis. Br J Clin Pharmacol. 2021 Jun;87(6):2589-2601. doi: 10.1111/bcp.14669. Epub 2020 Dec 16. PMID 33242339
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca